CLINICAL TRIAL: NCT02566161
Title: Parental Irradiation of Ukrainian Cleanup Workers and Evacuees and Germline Mutations in Their Offspring (Trio Study)
Status: Terminated | Type: Observational
Why Stopped: protocol qualifies as not human subjects research
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999915199; 15-C-N199
Record Dates: First submitted 2015-10-01; First posted 2015-10-02 (Estimated); Last update posted 2021-03-12 (Actual); Status verified 2020-07

CONDITIONS: Genetics
Keywords: Genetics; Genomics

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trio Cohort: families were from each of 5 exposure categories: A-father exposed, mother unexposed; B-mother exposed, father unexposed; C-both parents exposed; D-neither exposed; E-high dose emergency workers).

SUMMARY:
Data on transgenerational effects following nuclear accidents are important for understanding fully the consequences of parental exposure to ionizing radiation. Few studies to date have had adequate statistical power to detect effects of the magnitude expected based on animal data, and most have not been of low-dose, protracted exposures associated with nuclear accidents and their aftermath. Although, to date, scant use has been made of the new genomic technologies, in Chernobyl-exposed areas of Ukraine and Belarus, excess minisatellite mutations have been seen in children born after the accident. We propose a study of parent-child trios in which at least one parent was exposed to Chernobyl radiation as a clean-up worker (mean dose >=100 mGy) and/or evacuee from a contaminated area (mean >= 50mGy). The specific aims are to investigate the transgenerational and de novo mutation rates of the spectrum of genetic variants in trios, in particular looking at effects in children and mapping them to possible parental origin of the chromsome. Together with long-term collaborators at the Research Center for Radiation Medicine (RCRM) in Kiev, epidemiologic data will be collected for up to 450 trios of parents with preconceptional doses and their unexposed offspring. We will use state-of-the-art genomic technologies to characterize the landscape of the genomes of the trios to determine whether parental radiation exposure is associated with genetic mutations transmitted to the offspring, by examining de novo mutation rates, minisatellite mutations, copy number alterations, and variations in telomere length. The analysis will be conducted in peripheral blood and/or buccal samples (when blood is not available) from complete father-mother-child trios. Doses to the gonads from the time of the accident to the time of conception will be reconstructed for all parents using existing records supplemented by interview data.

Trio subjects will be selected from representative populations exposed to radiation from Chernobyl who are under active follow-up in the Clinico-Epidemiologic Registry at RCRM. To help identify specific effects of paternal and maternal radiation exposure, we will initially select sets of trio subjects in five categories: (1) exposed father, unexposed mother; (2) unexposed father, exposed mother; (3) both parents exposed; (4) both parents unexposed; and (5) a group of high dose emergency workers with acute radiation syndrome. All trio members will be invited to the RCRM outpatient clinic for collection of a 20 ml blood sample (or buccal cells for those who refuse phlebotomy). Both parents will be asked to complete a general questionnaire to obtain demographic and lifestyle data. Then one or both will complete detailed dosimetry questionnaires, based on forms used in previous collaborations with RCRM and administered by specially trained interviewers. Once 50 trios have been recruited (10 from each of the 5 exposure categories), we will conduct an interim evaluation of participation rates, sample collection and quality, and dose reconstruction in order to modify the protocol as needed. The analytical approach will be to correlate the extent, especially for de novo events of genetic alterations in the offspring with parental preconceptional radiation dose overall and by parental origin. The statistical power in relation to de novo mutations is very high, in excess of 90%, but somewhat lower for trends in minisatellite mutations. Study findings will contribute importantly to knowledge of the heritable effects of moderate- and low-dose radiation exposure in humans and to radiation risk projection. Eventually data from the Trio Study may be shared with the international community through dbGap.

DETAILED DESCRIPTION:
Data on transgenerational effects following nuclear accidents are important for understanding fully the consequences of parental exposure to ionizing radiation. Few studies to date have had adequate statistical power to detect effects of the magnitude expected based on animal data, and most have not been of low-dose, protracted exposures associated with nuclear accidents and their aftermath. Although, to date, scant use has been made of the new genomic technologies, in Chernobyl-exposed areas of Ukraine and Belarus, excess minisatellite mutations have been seen in children born after the accident. We propose a study of parent-child trios in which at least one parent was exposed to Chernobyl radiation as a clean-up worker (mean dose >=100 mGy) and/or evacuee from a contaminated area (mean >= 50mGy). The specific aims are to investigate the transgenerational and de novo mutation rates of the spectrum of genetic variants in trios, in particular looking at effects in children and mapping them to possible parental origin of the chromsome. Together with long-term collaborators at the Research Center for Radiation Medicine (RCRM) in Kiev, epidemiologic data will be collected for up to 450 trios of parents with preconceptional doses and their unexposed offspring. We will use state-of-the-art genomic technologies to characterize the landscape of the genomes of the trios to determine whether parental radiation exposure is associated with genetic mutations transmitted to the offspring, by examining de novo mutation rates, minisatellite mutations, copy number alterations, and variations in telomere length. The analysis will be conducted in peripheral blood and/or buccal samples (when blood is not available) from complete father-mother-child trios. Doses to the gonads from the time of the accident to the time of conception will be reconstructed for all parents using existing records supplemented by interview data.

Trio subjects will be selected from representative populations exposed to radiation from Chernobyl who are under active follow-up in the Clinico-Epidemiologic Registry at RCRM. To help identify specific effects of paternal and maternal radiation exposure, we will initially select sets of trio subjects in five categories: (1) exposed father, unexposed mother; (2) unexposed father, exposed mother; (3) both parents exposed; (4) both parents unexposed; and (5) a group of high dose emergency workers with acute radiation syndrome. All trio members will be invited to the RCRM outpatient clinic for collection of a 20 ml blood sample (or buccal cells for those who refuse phlebotomy). Both parents will be asked to complete a general questionnaire to obtain demographic and lifestyle data. Then one or both will complete detailed dosimetry questionnaires, based on forms used in previous collaborations with RCRM and administered by specially trained interviewers. Once 50 trios have been recruited (10 from each of the 5 exposure categories), we will conduct an interim evaluation of participation rates, sample collection and quality, and dose reconstruction in order to modify the protocol as needed. The analytical approach will be to correlate the extent, especially for de novo events of genetic alterations in the offspring with parental preconceptional radiation dose overall and by parental origin. The statistical power in relation to de novo mutations is very high, in excess of 90%, but somewhat lower for trends in minisatellite mutations. Study findings will contribute importantly to knowledge of the heritable effects of moderate- and low-dose radiation exposure in humans and to radiation risk projection. Eventually data from the Trio Study may be shared with the international community through dbGap.

ELIGIBILITY:
* INCLUSION CRITERIA:
* all parent-offspring trios/quartets selected from the group of approximately 450 trios with offspring born 42 or more weeks after the last significant parental Chernobyl-related exposure. ---The offspring can be of either sex
* Must be an adult

(age (Bullet) 18 years at interview);

* If more than one child is born to a given set of parents, the first and last such eligible siblings will be selected for participation, in the interests of maximizing the variation of time from last exposure to conception, also to maximize the signal (by including offspring closest in time to the exposure, with less likelihood of removal of damaged sperm/oocytes, and by including offspring furthest in time from the exposure, with less likelihood of direct exposure of the child, and maximizing cumulative parental preconception gonadal dose).
* Twins will be especially informative given the comparable exposures in utero and in early life. A high proportion of the trios/quartets currently reside in Kyiv. The majority of these trios/quartets have undergone regular medical examinations as a result of follow-up by the CER. Most of them are expected to be alive.

EXCLUSION CRITERIA:

* Those who cannot be located
* Those with offspring born within 42 weeks of the last significant Chernobyl-related exposure
* Those parents or offspring found to have cancer
* Those who refuse to participate in the study, or who do not provide informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Clinical-Epidemiological Registry (CER) of the RCRM will serve as the fundamental information source for the identification of potential trio subjects. The CER was established in 1992 for long-term extended active follow-up of representative populations exposed to ionizing radiation due to the Chernobyl nuclear power plant (ChNPP)accident, drawn from those listed in the State Chernobyl Registry. The study will include all parent-offspring trios/quartets selected from the group of approximately 450 trios with offspring born 42 or more weeks after the last significant parental Chernobyl-related exposure.
Sampling Method: Non-Probability Sample
Enrollment: 957 (Estimated)
Dates: Start 2015-10-01 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to investigate the association of parental preconceptual gonadal dose with genetic alterations in the offspring. | following sample collection
  Inherited genetic mutations

CONTACTS AND LOCATIONS:
Overall Officials: Amy Berrington, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Research Center for Radiation Medicine, Kiev, Ukraine

REFERENCES:
- [Background] Little MP, Goodhead DT, Bridges BA, Bouffler SD. Evidence relevant to untargeted and transgenerational effects in the offspring of irradiated parents. Mutat Res. 2013 Jul-Sep;753(1):50-67. doi: 10.1016/j.mrrev.2013.04.001. Epub 2013 May 4. PMID 23648355
- [Background] Dubrova YE, Grant G, Chumak AA, Stezhka VA, Karakasian AN. Elevated minisatellite mutation rate in the post-chernobyl families from ukraine. Am J Hum Genet. 2002 Oct;71(4):801-9. doi: 10.1086/342729. Epub 2002 Sep 11. PMID 12226793
- [Background] Bouffler SD, Bridges BA, Cooper DN, Dubrova Y, McMillan TJ, Thacker J, Wright EG, Waters R. Assessing radiation-associated mutational risk to the germline: repetitive DNA sequences as mutational targets and biomarkers. Radiat Res. 2006 Mar;165(3):249-68. doi: 10.1667/rr3506.1. PMID 16494513